CLINICAL TRIAL: NCT06027073
Title: Adding Biological Therapy to Asthmatic Patients on Allergen Immunotherapy to House Dust Mites
Brief Title: Biologics and Sublingual Immunotherapy
Acronym: BSIPL
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Centrum Medyczne Andrzej Bożek (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM-01966
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Asthma, Allergic
Keywords: IgE; asthma; omalizumab; immunotherapy
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: The randomization procedure with random selection will rely on computer-generated numbers using a computer program (Excel, version 14.2.0, 2020 Microsoft Corporation). The patients will be randomized into four groups 1:1:1:1 as follows:
  Group A: Xolair® Group B: Actair® Group C: Actair® and Xolair® Group D: Standard of Care (no interventional therapy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- omalizumab (Active Comparator): standard antiasthmatic therapy and omalizumab
  Interventions: Biological: omalizumab
- oral tablet HDM-immunotherapy (Active Comparator): standard antiasthmatic therapy and oral immunotherapy
  Interventions: Biological: omalizumab
- combi therapy (Active Comparator): standard antiasthmatic therapy and omalizumab, and oral immunotherapy
  Interventions: Biological: omalizumab
- control (No Intervention)

INTERVENTIONS:
Biological: omalizumab — adding omalizumab to anti asthmatic therapy
  Arms: combi therapy; omalizumab; oral tablet HDM-immunotherapy

SUMMARY:
Most current studies involve using a biological drug to increase the safety of allergen immunotherapy (AIT) especially in the treatment of food allergies, to avoid the risk of anaphylaxis. However, adding Xolair® to AIT may improve the therapy's effectiveness. There are still few observations on this topic, especially in patients with house dust mite (HDM)-driven asthma.

DETAILED DESCRIPTION:
Assess the effectiveness of combined therapy Actair® plus Xolair compared to monotherapy with Actair® or Xolair® or standard symptomatic therapy in patients with mild or moderate allergic asthma to HDM.

Treatment duration: 24 months Follow-up duration:12 months Total duration: 36 months (not including screening and randomization period) May 2024 - March 2028 Consisting of a 4 to 5 months screening phase (with 1 month observation period prior to randomization) a treatment phase of 24 months and post-treatment follow-up phase 12 months

ELIGIBILITY:
Inclusion Criteria:• >18 years old

* A total IgE between 30-700 IU/mL
* Moderate asthma with perennial symptoms confirmed as HDM-driven asthma based on medical history and positive nasal provocation tests, partially controlled asthma;
* FEV1 >70% at baseline;
* Positive skin prick test results for D. pteronyssinus, D. farinae

Exclusion Criteria:

* Sensitisation to other allergens with clinical signs not related to HDM
* Uncontrolled asthma,
* Other serious diseases or chronic unstable diseases
* Allergen immunotherapy during the past 5 years
* Contraindicating allergen immunotherapy and omalizumab treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of combined therapy : omalizumab+ immunotherapy | 3 years
  Daily dose of inhaled steroids (changes)

IPD SHARING:
Plan to Share IPD: No
by computer database registration

REFERENCES:
- [Derived] Batard T, Taille C, Guilleminault L, Bozek A, Floch VB, Pfaar O, Canonica WG, Akdis C, Shamji MH, Mascarell L. Allergen Immunotherapy for the Prevention and Treatment of Asthma. Clin Exp Allergy. 2025 Feb;55(2):111-141. doi: 10.1111/cea.14575. Epub 2024 Oct 4. PMID 39363801